CLINICAL TRIAL: NCT03079700
Title: Mucosal and Systemic Immune Modulation From Trichuris Suis in a Self-infected Individual
Brief Title: Immune Modulation From Trichuris Suis
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Christian Hvas, MD PhD, University of Aarhus
Other Study IDs: Trichuris suis
Record Dates: First submitted 2017-03-09; First posted 2017-03-14 (Actual); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Crohn Disease; Ulcerative Colitis; Intestinal Helminthiasis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Intestinal helminthiasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood cell and intestinal biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Trichuris suis eggs — Live eggs from swine whipworm, Trichuris suis

SUMMARY:
Mucosal immunology during helminth infection

DETAILED DESCRIPTION:
The present study investigates the effects of Trichuris suis on human mucosal and systemic immunity in a single self-infected individual.

ELIGIBILITY:
Inclusion Criteria:

* The included volunteer is a researcher within parasitology with main focus on Trichuris trichiura and Trichiura suis. He planned to infect himself and contacted our department with the purpose of being monitored during this infection for safety (medical supervision) and research reasons. The only clinical criterion for his inclusion in the study was that he was healthy.

Exclusion Criteria:

-

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A single healthy volunteer
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2012-08-01 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2012-12-31 (Actual)

PRIMARY OUTCOMES:
Faecal egg excretion | 15 weeks
  Weekly monitoring of fecal egg counts by microscopy

SECONDARY OUTCOMES:
Mucosal T cell associated cytokines | 15 weeks
  Biopsy sampling during established infection
Systemic immune parameters (eosinophilia, Subtypes of circulating T cells) | 15 weeks
  Blood samples every week
Adverse events | 15 weeks
  Clinical evaluation every week

IPD SHARING:
Plan to Share IPD: No